CLINICAL TRIAL: NCT00462774
Title: Evaluierung Eines Therapiemodells Der Autologen Knochenmark-Transplantation Bei Herzerkrankungen Mit Besonderem Schwerpunkt Der Prüfung Verschiedener Progenitorzellen
Brief Title: Bypass Surgery and CD133 Marrow Cell Injection for Treatment of Ischemic Heart Failure
Acronym: Cardio133
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: German Heart Institute (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHZB/CARDIO133/2007/1
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease With Need for Bypass Surgery; Myocardial Ischemia, Angina Pectoris; Congestive Heart Failure; Previous Myocardial Infarction
Keywords: Myocardial infarction; Heart failure; Cell therapy; Bone marrow; CD133; Bypass surgery; Stem cells
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Heart Failure; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Intramyocardial injection of autologous CD133+ marrow cells

SUMMARY:
Cell transplantation for treatment of heart failure is a novel field of translational research that offers the perspective of developing curative approaches by regenerating or "rejuvenating" lost and/or diseased myocardium and inducing growth of new blood vessels. Based on the safety and preliminary efficacy testing in previous trials, a stringent efficacy testing will be performed in this study. Sixty patients who had myocardial infarction in the past and now need bypass surgery for ongoing coronary artery disease will undergo either bypass surgery and placebo treatment or bypass surgery and injection of CD133 bone marrow cells directly in the heart muscle. The study will be fully blinded, i.e. neither the patient nor the surgeon knows what substance is injected (placebo or cell product). Patients will be followed for 6 months and various heart function measurements will be performed.

DETAILED DESCRIPTION:
Beginning in 2001, a phase-1 equivalent feasibility and safety evaluation of intramyocardial injection of autologous CD133+ bone marrow cells during elective CABG surgery was conducted at Rostock University. No procedure-related adverse events were observed and there was some improvement of myocardial contractility and perfusion. It was decided to proceed with a controlled efficacy testing, comparing the outcome of standard CABG surgery with that after CABG and CD133+ cell injection. The results of that study indicate that the additional cell injection yields a better left ventricular contractility than CABG alone (LVEF = 47.1±8% vs. 41.3±9% at 6 months). Although this result is encouraging, the trial had several limitations that hamper interpretation of the data. Most notably, no sham-injection of placebo material was performed in the control group, and standard 2D echocardiography served as the only measurement of global LV contractility. A more stringent efficacy testing is needed before large-scale clinical multicenter trials are justified.

Therefore, a prospective, full blinded, randomized, and placebo-controlled trial will be conducted at Deutsches Herzzentrum Berlin Berlin (DHZB), employing current state-of-the art measurement of global and regional LV contractility by cardiac MRI. The following hypothesis will be tested: "Patients who undergo CABG & CD133+ cell injection do not have a higher LV ejection fraction than patient who undergo CABG alone, measured 6 months after the operation". A power analysis based on the previous trial results indicated that 29 patients per group need to be enrolled so as to reject the null-hypothesis with sufficient statistical power. A total of 60 patients will therefore be enrolled in the study and will be randomized to undergo either CABG surgery and injection of placebo or in conjunction with intramyocardial injection of autologous CD133+ enriched bone marrow cells. Bone marrow will be harvested one day prior to surgery and a CD133-enriched cell product (or placebo) will be prepared on-campus. The following day, bypass surgery will be performed and the study substance will be injected in the border zone of the infarcted myocardium. Random allocation will be performed in the cell production facility, so that neither the patient nor the surgeon nor any of the persons involved in follow-up examinations will know whether the cell product or placebo was administered. The primary outcome parameter (LVEF at 6 months) will be measured by cardiac MRI, and secondary outcome parameters include myocardial perfusion, exercise capacity, and quality-of-life assessment.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease with indication for CABG surgery
* Reduced global left ventricular ejection fraction by transthoracic echocardiography at rest (EF ≤ 35%)
* Presence of a localized akinetic/hypokinetic/hypoperfused area of LV myocardium for defining the target area
* Informed consent of the patient
* Age > 18 years

Exclusion Criteria:

* Emergency operation
* Presence of aortic valve disease requiring concomitant valve replacement
* Debilitating other disease: Degenerative neurologic disorders, psychiatric disease, terminal renal failure requiring dialysis, previous organ transplantation, active malignant neoplasia
* History of ventricular arrhythmia (≥ Lown III)
* Impaired ability to comprehend the study information
* Absent informed written consent
* Apparent infection (CRP ≥ 20 mg/L, fever (≥38.5° C)
* Acute myocardial infarction
* contraindication for MRI assessment
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction at rest, measured six months postoperatively, measured by MRI

SECONDARY OUTCOMES:
Change in LVEF compared with preoperatively and early postoperatively
Regional contractility in the AOI
Physical exercise capacity determined by 6 minute walk test
Perfusion in the AOI
Change in LV dimensions
NYHA and CCS class
Minnesota Living with Heart Failure Score
Death, myocardial infarction, or need for reintervention during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Roland Hetzer, MD, PhD, Study Director — German Heart Institute; Boris Nasseri, MD, Principal Investigator — German Heart Institute; Christof Stamm, MD, Principal Investigator — German Heart Institute
Locations (1):
- Deutsches Herzzentrum Berlin, Berlin, Germany

REFERENCES:
- [Background] Stamm C, Westphal B, Kleine HD, Petzsch M, Kittner C, Klinge H, Schumichen C, Nienaber CA, Freund M, Steinhoff G. Autologous bone-marrow stem-cell transplantation for myocardial regeneration. Lancet. 2003 Jan 4;361(9351):45-6. doi: 10.1016/S0140-6736(03)12110-1. PMID 12517467
- [Background] Stamm C, Kleine HD, Choi YH, Dunkelmann S, Lauffs JA, Lorenzen B, David A, Liebold A, Nienaber C, Zurakowski D, Freund M, Steinhoff G. Intramyocardial delivery of CD133+ bone marrow cells and coronary artery bypass grafting for chronic ischemic heart disease: safety and efficacy studies. J Thorac Cardiovasc Surg. 2007 Mar;133(3):717-25. doi: 10.1016/j.jtcvs.2006.08.077. Epub 2007 Feb 1. PMID 17320570
- [Derived] Nasseri BA, Ebell W, Dandel M, Kukucka M, Gebker R, Doltra A, Knosalla C, Choi YH, Hetzer R, Stamm C. Autologous CD133+ bone marrow cells and bypass grafting for regeneration of ischaemic myocardium: the Cardio133 trial. Eur Heart J. 2014 May 14;35(19):1263-74. doi: 10.1093/eurheartj/ehu007. Epub 2014 Feb 3. PMID 24497345